CLINICAL TRIAL: NCT00500500
Title: Effect of EGb 761® on the Ratio of the Isoforms of the Protein Precursor of Beta Amyloid Platelets on Patients With Mild to Moderate Alzheimer's Disease. A Phase II, Randomised, Double-blind Trial, on Parallel Groups Versus Placebo.
Brief Title: Effect of EGb 761® on Patients With Mild to Moderate Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inability to recruit sufficient number of patients
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2-29-00240-127
Record Dates: First submitted 2007-07-11; First posted 2007-07-12 (Estimated); Last update posted 2023-06-26 (Actual); Status verified 2013-10

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Ginkgo biloba extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- EGb 761® (Tanakan®) (Experimental): EGb 761® (Tanakan®)
  Interventions: Drug: EGb 761® (Tanakan®)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: EGb 761® (Tanakan®)

INTERVENTIONS:
Drug: EGb 761® (Tanakan®)

SUMMARY:
The aim of this study is to measure the effect of EGb 761® versus placebo on the ratio of the isoform of the protein precursor of beta amyloid platelets, in patients with mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* female or male of 50 to 85 years old with a care giver
* Mini Mental Status (MMS) test between 16 to 26 inclusive
* Clinical Dementia Rating (CDR) test inferior or equal to 1
* National Institute of Neurological and Communicative Disorders and Stroke / Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) test positive for an Alzheimer's disease
* Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM IV) test positive for dementia

Exclusion Criteria:

* patient already treated by medicines which could interfere with the study
* low level of vitamin B12 and folate which are considered as clinically relevant
* clinically relevant pathologies (eg: pulmonary illness, cardiovascular illness; evolutive cancer, neurological illness, blood illness….)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Effect of EGb 761® on the ratio of the isoform of the protein precursor of beta amyloid platelets. | Every visit

SECONDARY OUTCOMES:
Efficacy of EGb 761® on the cognitive functions and safety of EGb 761® at a dosage of 240 mg per day | Every visit

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Ipsen
Locations (1):
- Hôpital La Timone, Marseille, France